CLINICAL TRIAL: NCT04790019
Title: The Effects of Short-term Low Energy Availability and Low Repetition High Impact Jumping on Markers of Bone Formation and Resorption in Young Females
Brief Title: The Effects of Low Energy Availability and High Impact Jumping on Markers of Bone (re)Modelling in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Katherine Brooke-Wavell, Principle Investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R20-P052
Record Dates: First submitted 2020-10-02; First posted 2021-03-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Bone Resorption; Bone Atrophy; Energy Supply; Deficiency; Female Athlete Triad; Relative Energy Deficiency in Sport
Keywords: Low energy availability; Energy restriction; Bone (re)modelling; Bone metabolism; High impact exercise
MeSH Terms: conditions — Bone Resorption; Female Athlete Triad Syndrome; Relative Energy Deficiency in Sport

STUDY DESIGN:
Intervention Model Description: All participants will complete the control condition and one of two experimental conditions in a randomized and counterbalanced crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low energy availability (Experimental): Intervention involves three of dietary energy restriction providing 15 kilo-calories per kilogram of fat-free mass per day.
  Interventions: Behavioral: Low energy availability
- Low energy availability and high impact jumping (Experimental): Intervention involves three days of dietary energy restriction providing 15 kilo-calories per kilogram of fat-free mass per day and brief high impact jumping exercise performed daily in the morning and in the evening.
  Interventions: Behavioral: Low energy availability; Behavioral: High impact jumping

INTERVENTIONS:
Behavioral: Low energy availability — Participants will be provided with food to eat every day and will not be permitted to consume any other calorie containing foods or beverages. This amount of energy contained within the food provided will be one third of that contained in the food provided in the control condition (45 kilo-calories per kilogram of fat-free mass per day) and will be standardized between and within participants for carbohydrate, protein and fat composition.
  Other Names: Energy restriction
Behavioral: High impact jumping — Participants will perform a brief session of high impact jumping every morning (10 maximum effort vertical counter-movement jumps, and 5 maximum effort lateral drop jumps in each direction) and a similar session of high impact jumping every evening (20 maximum effort vertical counter-movement jumps).
  Arms: Low energy availability and high impact jumping

SUMMARY:
Osteoporosis is worldwide health epidemic categorized by poor bone health, primarily diagnosed by low bone mineral density, and costs healthcare systems billions every year. Athletes and exercising people who expend large amounts of energy in physical activity, or restrict diet in order to lose weight, are at risk of low energy availability. This is when an individual fails to match their exercise energy demand with a appropriate dietary intake in order to maintain optimal physiological function; which can lead to low bone mineral density, osteoporosis both early and later in life and an increased risk of injury. Runners are particularly susceptible to stress fracture in response to low energy availability due to repetitive ground impact. Research shows that as little as five days low energy availability significantly reduces bone formation, and significantly increases bone resorption, in physically active women. The ideal solution is to restore energy availability; however, this is often very difficult during periods of intense training and conflicts with the goal of weight loss. Therefore, there is a need to develop an alternative tool to protect bone health. It is critical that any exercise intervention does not further reduce energy availability as previous research shows that this accelerates bone loss rather than prevents it. Low repetition high impact jumping exercise is highly beneficial to bone health and has been shown to improve bone structure when used as a long-term intervention in energy replete states. It takes very little time to complete and uses a very small amount of energy. However, no study to date has examined the effects of such an intervention during low energy availability. The current study will investigate whether low repetition high impact jumping prevents or reduces the reduction in bone formation and the increase in bone resorption experienced during five days of low energy availability and findings will have implications on athletic and recreational training recommendations in order to protect bone health.

DETAILED DESCRIPTION:
Participants will complete two four-day experimental conditions within the first seven days of two separate menstrual cycles. These will be preceded by a four-day baseline assessment period. There are three experimental conditions in total: control (CON), low energy availability (LEA) and low energy availability and high impact jumping (LEA+J). Participants will be randomly allocated to complete the control condition and either the LEA or LEA+J condition. The order in which the two conditions are completed will be randomized and counterbalanced. In total, fifteen laboratory visits will be required per participant:

Baseline assessment (four days and one visit):

Visit 1:

Participants will come to the laboratory to complete the informed consent procedure on day 1, once they have had at least 24 hours to consider the participant information sheet. Providing informed consent is given, participants will complete three questionnaires (a health screen, the Low Energy Availability in Females Questionnaire and the International Physical Activity Questionnaire) which include questions regarding their medical and injury history, dietary habits, menstrual cycle and physical activity habits. They will then have their height and weight taken. Provided the responses and measures confirm that the participant meets the inclusion and exclusion criteria, they will then undergo familiarization of resting metabolic rate assessment where they will lay supine in a dimly lit room whilst expired gas is collected via a mouthpiece. During familiarization the researcher will check for signs of hyperventilation. Following that, the participants will be familiarized with a jumping exercise routine if the participant is randomized into the group that will be performing this routine during an experimental condition. Finally, the participant will be asked to complete an incremental exercise test to volitional exhaustion on a treadmill whilst expired gas is collected and analysed using a metabolic cart, and heart rate and rating of perceived exertion are taken, as a measure of aerobic fitness.

For the following three days (2, 3 and 4), participants will be instructed to self-report weighed energy intake using a set of scales provided and a food diary according to the instructions on the diary itself which the researcher will read through with the participant. They will be asked to eat according to their usual dietary habits and return it electronically at the end of day 4, or during a subsequent visit. Participants will also be provided with a tri-axial accelerometer (Actigraph GT3X+) device and instructed to wear it around the waist for the entirety of days 2, 3 or 4 (apart from when bathing and washing). They will be not required to visit the laboratory on days 2, 3 or 4.

Experimental conditions (four days and four visits, per condition):

The following will outline the experimental protocol assuming the participant is completing the LEA+J condition followed by the CON condition, and end with a description of how the protocol differs should they be randomly allocated to complete the LEA condition as opposed to the LEA+J, condition. Participants will be required to refrain from exercise which is not part of the study for the entirety of all experimental conditions.

LEA+J condition:

Participants will be required to notify the research team at the onset of their next menses and will commence the experimental condition the following day, or the day after that if the participant is not able to do what is required of them the following day. From the first until the last day of each condition, participants will be required to wear the Actigraph device at all times apart from when bathing and washing. Participants will be instructed to record their diet during day 1, as they did during days 2, 3 and 4 of the baseline condition, and will be asked to eat according to their usual dietary habits but instructed to make choices that they will be able to replicate ahead of each subsequent experimental condition. They will not be permitted to drink caffeine or alcohol.

Visit 1:

Participants will be required to collect their final meal on day 1 from the laboratory and will be instructed to eat it at exactly 20:00. They will complete the Pittsburgh Sleep Quality Index (PSQI; a questionnaire regarding sleep habits and quality during the last month). They will also be instructed to refrain from any other food or drink, other than water, for the rest of the evening. Participants will be provided with a self-report water intake record sheet and water bottle from which to drink and instructed to report daily water intake from the start of day 2 until the end of the condition. They will also be provided with a small container suitable to collect a urine sample upon waking the following morning. Participants will be instructed to bring the sample with them to the laboratory, where it will be analysed and disposed of immediately.

Visit 2:

On day 2 of the first condition, participants will be required to arrive at the laboratory between 06:00-09:00 without eating breakfast or ingesting caffeine for at least 18 hours prior. The participant will be asked to travel by car or by public transport and restrict walking distance as much as possible. Weight and body composition will be taken in shorts and underwear using scales and bio-electrical impedance. The investigators will then perform a resting metabolic rate assessment and a series of cardiovascular measures using pressure cuffs, tonometry and electrocardiography. A venous blood sample will be split into plasma and serum separation Vacutainers from the arm by a phlebotomy trained researcher using standard venepuncture methods. The participants will then be instructed to complete a brief high impact jumping exercise routine on a Kistler force platform with demonstrations by the researcher and continued feedback to maintain optimum form. All jumps will be performed barefoot. The investigators will then provide a breakfast to consume in the laboratory along with a multivitamin multi-mineral tablet. The food the participants are required to eat for the rest of the day will be packed into a cool box to take away and the participants will not be permitted to consume anything which is not provided within the cool box, other than "calorie-free" drinks (black coffee, black tea, green tea, etc.). The participants will be instructed to perform a similar jump routine at home at least 8 hours after the morning jump routine. All jumps will be performed barefoot.

Visits 3 and 4:

On days 3 and 4, participants will be required to arrive at the laboratory between 06:00-09:00 without eating breakfast. Participants will return any uneaten food from the previous day and report any items consumed (other than "calorie-free" drinks) that were not part of the cool box provided. The participants will complete the morning jump routine and have their prescribed breakfast with multivitamin and multi-mineral tablet at the laboratory, before leaving with the rest of their food for that day packed in a cool box. The participants will not be permitted to consume anything which is not provided within the cool box, other than "calorie-free" drinks. The participants will be instructed to complete the evening jump routine - as on day 2.

During day 4, participants will only be permitted to drink water and will be instructed to consume their final meal at 20:00 and refrain from any other food or drink (other than water) for the rest of the evening. At the end of day 6, the participants will also be provided with a small container suitable to collect a urine sample upon waking the following morning. Participants will be instructed to bring the sample with them to the laboratory, where it will be analysed and disposed of immediately.

Visit 5:

On day 5, participants will repeat the same process as on day 2, except will be required to arrive at the laboratory at the exact same time rather than anywhere between 06:00 - 09:00 and they will not complete the morning or evening jump routines, the PSQI or be given breakfast, a multivitamin multi-mineral tablet nor food to take away.

Participants will be provided with an ovulatory test kit to take away and use once per day (urinate on a stick as per a pregnancy test) for up to 8 days in the middle of the menstrual cycle. Once a positive test is observed the participants will report this to the research team and if no positive is reported within 8 days this will also be reported to the research team.

CON condition:

Visits 1-5:

Participants will again be required to notify the research team at the onset of the next menses (following the end of the LEA+J condition) and will commence the CON condition the following day, or the day after that if the participant is not able to do what is required of them the following day. The same procedure as in the LEA+J condition will be repeated, however, rather than recording their diet during day 1, participants will be instructed to repeat what was previously recorded. Also, the total energy intake in the food provided in the LEA+J condition will be a third of that provided in the CON condition and participants will not take a multivitamin multi-mineral tablet or be required to perform morning or evening jump routines.

How will the protocol differ for participants completing the LEA condition?

The procedure for the LEA condition is the same as in the LEA+J condition, however, participants will not be required to perform morning or evening jump routines.

ELIGIBILITY:
To take part in this study, the following inclusion criteria must be met:

* Menstrual cycles that are between 21 - 35 days in length for at least the previous three cycles
* Regular length of menstrual cycle (less than six days difference between cycles) for at least the previous three cycles
* Body mass index between 18.5 - 30 kg.m squared
* Weight stable for the past three months and not currently dieting

Participants will not be able to take part in this study if any of the following exclusion criteria are met:

* Smoker
* Pregnant
* Vegan
* Have used hormonal contraception at any point within the previous three months
* Regularly engage in >3 vigorous, or >5 moderate, exercise sessions a week
* Compete regularly in a high or multi-directional impact sport at national level or higher
* Have sustained a bone injury within the previous twelve months
* Have sustained any injury within the past six months that restricted their ability to exercise
* Taken hormone replacement therapy (HRT) at any point during the past three months
* Have been previously diagnosed with an eating disorder
* Have taken any medications (other than vitamin or mineral supplements) known to effect bone metabolism within the previous three months (e.g. glucocorticoids, anticonvulsants or anabolic steroids)
* Have previously been diagnosed with a medical condition known to impact bone health (e.g. hypothyroidism, hyperthyroidism, diabetes mellitus, hypercortisolism and renal or gastrointestinal disease)
* Have previously been diagnosed with a pathology known to impact menstrual function (e.g. primary ovarian insufficiency, hyperprolactinemia, thyroid dysfunction, polycystic ovarian syndrome and any other conditions of androgen excess)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in blood pro-peptide of type 1 collagen (P1NP) concentration | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  P1NP is a marker of bone resorption and it will be measured during the fasted state
Change in blood β-carboxyl-terminal cross-linked telopeptide of type 1 collagen (β-CTx) concentration | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  β-CTx is a marker of bone formation and it will be measured during the fasted state

SECONDARY OUTCOMES:
Change in blood 17β-oestradiol concentration | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  17β-oestradiol is a reproductive hormone that fluctuates during the menstrual cycle and is involved in the regulation of bone resorption
Change in blood triiodothyronine (T3) concentration | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  T3 is a thyroid hormone that has previously been shown to decrease in response to low energy availability has been proposed as a useful marker of low energy availability
Change in blood β-hydroxybutyrate (β-OHB) concentration | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  β-OHB is a ketone body produced during periods of energy and/or carbohydrate restriction
Change in blood calcium concentration | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  Calcium is a micro-nutrient involved in the regulation of bone (re)modelling and may change in response to low energy availability
Change in blood magnesium concentration | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  Magnesium is a micro-nutrient involved in the regulation of bone (re)modelling and may change in response to low energy availability
Change in blood phosphorus concentration | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  Phosphorus is a micro-nutrient involved in the regulation of bone (re)modelling and may change in response to low energy availability
Change in resting metabolic rate (RMR) | From the morning of the first day of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  This is amount of energy used by the body at rest and is measured via indirect calorimetry compared to RMR predicted using previously validated equations. It has been proposed that a ratio of <0.9 may be used as a surrogate marker of energy deficiency
Change in ratio of measured:predicted resting metabolic rate (RMR) | From the morning of the first day of dietary provision to the same time on the morning following the final day of dietary provision (five days later), in each condition
  This is the ratio of RMR measured via indirect calorimetry compared to RMR predicted using previously validated equations. It has been proposed that a ratio of <0.9 may be used as a surrogate marker of energy deficiency
Change in blood plasma volume (estimated using haemoglobin concentration and haematocrit) | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  Plasma volume is a measure of the proportion of blood that is made up of plasma. It has been shown to change in response to low energy availability and may influence the concentrations of primary measures independent of low energy availability, per se.
Change in heart rate variability | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  It has been proposed that low energy availability impairs cardiovascular function and heart rate variability is a measure of the variation in time between each heart beat
Change in the spectral density of heart rate variability in low and high frequency bands | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  It has been proposed that low energy availability impairs cardiovascular function and spectral analysis of heart rate variability provides information on the function of sympathetic and parasympathetic regulation of heart rate
Change in aortic stiffness | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  It has been proposed that low energy availability impairs cardiovascular function and aortic stiffness is estimated via measurement of arterial stiffness at the wrist
Change in forearm resting blood flow | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  It has been proposed that low energy availability impairs cardiovascular function and forearm blood flow is a marker of cardiovascular function that can be measured using plethysmography
Change in forearm peak blood flow | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  It has been proposed that low energy availability impairs cardiovascular function and peak forearm blood flow is a marker of cardiovascular function that can be measured using plethysmography
Change in body weight | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  Body weight could be expected to decrease in response to caloric restriction and will therefore be measured and can be used to indicate adherence to dietary provision
Change in fat-free mass | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  Fat-free mass could be expected to decrease in response to caloric restriction and will therefore be measured and can be used to indicate adherence to dietary provision
Change in baroreflex sensitivity | of dietary provision to the same time on the morning following the final day of dietary provision (three days later), in each condition
  It has been proposed that low energy availability impairs cardiovascular function and baroreflex sensitivity is a marker of the functionality of the system of cross-talk between cardiac control and blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Blagrove, PhD, Principal Investigator — Loughborough University; Emma O'Donnell, PhD, Study Director — Loughborough University; Katherine SF Brooke-Wavell, PhD, Study Director — Loughborough University
Locations (1):
- Mark Hutson, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No